CLINICAL TRIAL: NCT06067789
Title: Anesthesia for Lower Limb Revascularization to Optimize Functional ouTcomes
Brief Title: The ALOFT Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Ottawa Hospital Academic Medical Association (Other); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTO-TBD
Record Dates: First submitted 2023-09-14; First posted 2023-10-05 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Vascular Diseases; Peripheral Artery Disease; Surgery
MeSH Terms: conditions — Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Group allocation will not be indicated in data analyzed by the outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention arm participants will be allocated to neuraxial anesthesia. The specific approach (spinal, epidural, or combined spinal and epidural) will be at the discretion of the treating anesthesiologist, as the underlying physiologic mechanisms and impacts are similar for both approaches. Allowing clinician discretion will reflect routine standard of care practice and support generalizability. Specific choice of neuraxial anesthetic medications, doses, and adjuncts will also be at the discretion of the attending anesthesiologist, supporting pragmatism. While existing randomized data do not suggest that the sedation level during neuraxial anesthesia leads to differences in outcomes, providers will be requested to maintain sedation at or below a 3 on the Observer's Assessment of Alertness/Sedation scale (OAAS; mild to moderate sedation consistent to responding to verbal stimuli), the same approach used in a recent large pragmatic trial of anesthesia in hip fracture patients.
  Interventions: Procedure: neuraxial anesthesia
- Control (No Intervention): Control group participants will be allocated to general anesthesia. Choice of anesthetic medications and doses will be at the discretion of each anesthesiologist as per routine standard of care, again supporting conduct of a pragmatic and generalizable trial. Similarly, choice of airway management strategies and anesthetic depth will also be based on patient and provider preference, as a recent large randomized trial demonstrates that anesthetic depth is not causally linked to risk of morbidity or mortality after surgery. Details of general anesthesia management and medications will be collected for all patients.

INTERVENTIONS:
Procedure: neuraxial anesthesia — Intervention arm participants will be allocated to neuraxial anesthesia.
  Arms: Intervention

SUMMARY:
The ALOFT Pilot Trial will evaluate three pragmatic elements (recruitment, adherence, and follow-up) of neuraxial versus general anesthesia for lower limb revascularization surgery that are necessary to support a successful, large-scale evaluation. We will concurrently use implementation science methodology to further refine processes for the larger trial.

The future full ALOFT trial will be designed to evaluate the comparative effectiveness of two different anesthesia types for improving outcomes.

DETAILED DESCRIPTION:
Background: Despite promising evidence suggesting benefit from neuraxial anesthesia for lower limb revascularization surgery, our data demonstrate that use of neuraxial anesthesia varies 6-fold between Canadian hospitals and is decreasing over time. Currently available evidence is largely observational. Only data from a multicenter, randomized trial of anesthesia type for lower limb revascularization surgery, powered for patient-reported outcomes and designed with patient and knowledge user partners, will provide the high-certainty evidence of the possible benefits of neuraxial anesthesia. Therefore, we are designing the Anesthesia for Lower limb revascularization to Optimize Functional ouTcomes (ALOFT) Trial to address this important question. Prior to conducting this full trial, the feasibility of the trial protocol must be demonstrated using a multicenter pilot design.

Overarching Aim: The ALOFT Pilot Trial will evaluate three pragmatic elements (recruitment, adherence, and follow-up) of neuraxial versus general anesthesia for lower limb revascularization surgery that are necessary to support a successful, large-scale evaluation.

Methods:

Design, setting and participants:

The ALOFT Pilot Trial is an assessor blinded, multicenter, individual patient, parallel-arm randomized controlled trial.

People => 18 years with a planned lower limb revascularization surgical procedure (on an elective or urgent basis): infrainguinal arterial bypass, femoral endarterectomy, patch angioplasty will be included.

Intervention: The intervention arm participants will be allocated to neuraxial anesthesia. The specific approach (spinal, epidural, or combined spinal and epidural) will be at the discretion of the treating anesthesiologist, as the underlying physiologic mechanisms and impacts are similar for both approaches.

Outcomes and sample size: Primary outcome is monthly recruitment. Secondary outcomes are intervention adherence, retention, and elicitation of patient, clinician and researcher-identified barriers. Our pilot trial sample size estimate is informed by a power calculation for the future full-scale trial. In the future trial, a sample of 778 (389/arm) will provide 90% power using ANCOVA to detect the 5% minimally important between group difference in the continuous WHODAS score assuming a common standard deviation of 20 and a correlation with baseline of 0.4 (as observed in our previous work4) as well as accounting for up to 10% attrition and up to 10% cross-over. For the pilot trial, a sample size of 90 directly links to our 3 feasibility outcomes.

Expertise: Our team features multidisciplinary clinical and methodological experts, nationally representative knowledge users and patient representatives.

Expected outcomes: Our objective is for results of the planned full trial to change practice in caring for lower limb revascularization surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Planned lower limb revascularization surgical procedure (on an elective or urgent basis): infrainguinal arterial bypass, femoral endarterectomy, patch angioplasty
3. Able to access a telephone for postoperative follow-up

Exclusion Criteria:

1. Absolute contraindications to neuraxial anesthesia: impaired coagulation state (due to intrinsic, congenital or extrinsic (i.e., anticoagulant not held for guideline recommended period based on the American Society of Regional Anesthesia recommendations) factors), infection at the needle insertion point, increased intracranial pressure or intracranial mass, uncorrected hypovolemia or hypotension (systolic blood pressure <90 mmHg), severe uncorrected aortic stenosis)
2. Traumatic arterial injuries as an indication for surgery
3. Multiple sclerosis or demyelinating central nervous system conditions
4. Known malignant hyperthermia or who require a malignant hyperthermia trigger-free anesthetic
5. Pregnancy
6. Prior enrollment in this study, or participating in another interventional trial that could interfere with interpretation of data for either study (may be acceptable if unrelated interventions/outcomes and study PIs mutually agree in writing to co-enrollment)
7. Determination by the surgeon, anesthesiologist, or other clinician, that the patient would not be suitable for randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Monthly recruitment | 2 years
  Monthly recruitment of >=2 participants per center means that the full trial should be feasible

SECONDARY OUTCOMES:
Intervention adherence | 1 day
  >=90% of participants were treated with allocated randomization arm to minimize the risk of contamination bias
Retention | 30 days
  >=90% of participants at the patient-reported primary outcome point of 30-days after surgery should minimize attrition bias in the definitive trial's primary outcome data
Elicitation of patient, clinician and researcher-identified barriers and facilitators | 30 days, 120 days
  For study participants, at 30-day follow-up, a survey will be administered focusing on the acts of enrolling and being followed up in the trial. For research team members, a survey focused on the acts of participant recruitment and study support will be done once per site for all researchers, inclusive of clinician researchers and research staff, at approximately 3-4 months after study launch at their site.

OTHER OUTCOMES:
Rate of suspected spinal cord hematomas or infections | 1 year
  Measured by the number of participants requiring spinal imaging
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 30 days, 90 days, 1 year
  Patient-reported disability scale that assesses limitations in six major life domains (cognition, mobility, self-care, social interaction, life activities, participation in society). Each questionnaire item is scored on a Likert scale ranging from 0 to 4. The sum of the responses is the WHODAS Disability Score (range: 0 to 48), which is expressed as a percentage of the maximum possible score. People who die prior to follow up are assigned a score of 100% (completely disabled).
EuroQol Health-related quality of life (EQ-5D-5L) | 30 days, 90 days, 1 year
  Well-validated instrument with Canadian valuation statistics and national implementation used to measure health-related quality of life at baseline, 30, 90, and 365 days after surgery and to inform incremental cost per quality-adjusted life year gained. Each item in the EQ-5D-5L has five levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5).
Pain Score | up to 3 days, 30 days, 90 days, 1 year
  A numeric rating scale pain score (worst and average) will be collected at each prospective assessment point. Likert scale from 0-10 will be used where 0=No Pain At All and 10=Worst Possible Pain.
Satisfaction with anesthesic technique: 'Likelihood to recommend', reflecting on a 10-point scale their likelihood to recommend their anesthetic technique to a future patient having the same surgery | up to 3 days
  At the first in-hospital follow up patients will complete the 'Likelihood to recommend' question, where they will report a score from 0=Not at all likely to recommend to 10=Very likely to recommend.
Quality of Recovery Score: How well the patient feels they have recovered from their anesthetic and operation | up to 3 days
  At the first in-hospital follow up patients will answer 15 questions regarding how they have been feeling in the last 24 hours and will score each question on a Likert scale. The scoring for the first 10 questions goes from 0 to 10, where 0=they experience the issue none of the time [poor] and 10=they experience the issue all of the time [excellent]. For the last 5 questions the score goes from 10 to 0, where 10=they experience this symptom none of the time [excellent] and 0=all of the time [poor]. Results are totalled to provide an overall score for the 15 questions
Delirium | 1 month
  Using the validated chart review tool, Chart-based Delirium Identification Instrument
Complications | 1 month
  The validated and widely used Post-Operative Morbidity Survey (POMS) will be used to identify complications from the medical record; severity will be assessed using the Clavien-Dindo classification. At time of discharge, participants will also be administered a patient-reported version of the POMS tool.
Index hospitalization | 1 month
  Length of stay post-surgery and discharge disposition post-surgery
Major adverse limb events | 30 days, 90 days, 1 year
  Collected from medical records and by telephone follow up using Society of Vascular Surgery criteria
Days at home | 30 days
  In the 30-days after surgery, is a validated patient-centered, outcome that can be ascertained from routinely collected data
Readmission | up to 1 year
  Time to first, and count of any, acute hospitalization
Emergency department visits | up to 1 year
  Time to first, and count of any emergency department visits
Survival | up to 1 year
  All cause deaths and survival time after surgery will be captured from medical records and by telephone follow up.
Healthy system costs | up to 1 year
  A validated patient-level costing algorithm will be used to capture all health system costs accrued after surgery
Rate of spinal hematomas or infections | 1 year
  Measured by the number of participants requiring surgery to decompress or evacuate a spinal hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Daniel McIsaac, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including data dictionaries, will be available. This includes individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The Study Protocol, Statistical Analysis Plan and Informed Consent Form will also be made available. Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data. Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.
Supporting Information: SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.